CLINICAL TRIAL: NCT02215057
Title: Evaluation of Topical Anesthesia Alone Versus Combined With Intracameral Lidocaine 1% in Patients Undergoing Implantable Collamer Lens (ICL) Procedure
Brief Title: Evaluation of Topical Anesthesia Alone Versus Combined With Intracameral LIdocaine 1%
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1479
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Other Iris and Ciliary Body Disorders
Keywords: topical anesthesia; intracameral lidocaine; implantable collamer lens
MeSH Terms: interventions — Anesthesia; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Experimental): topical anesthetic drops patients were prepared for bilateral ICL/TICL procedure on the same day.Group I (1 eye) received topical anesthetic drops
  Interventions: Drug: topical anesthesia
- Group 1 (Experimental): received topical anesthesia plus intracameral lidocaine 1% topical anesthesia plus intracameral lidocaine 1%'
  Interventions: Drug: topical anesthesia; Drug: topical anesthesia plus intracameral lidocaine 1%

INTERVENTIONS:
Drug: topical anesthesia — topical anesthetic drops and Group 2
  Other Names: LOCAL ANESTHESIA
Drug: topical anesthesia plus intracameral lidocaine 1% — received topical anesthesia plus intracameral lidocaine 1%
  Other Names: received topical anesthesia plus intracameral lidocaine 1%
  Arms: Group 1

SUMMARY:
General anesthesia may be non preferable in many patients undergoing Phakic IOL surgery, as most of the surgeries take 5-10 minutes at maximum.Traditionally, retrobulbar injections were performed deep into the orbit, but it is now accepted that peribulbar injections using shorter needles are safer. In the last few years, continuing concern over the rare but serious complications of sharp needle blocks has led to increasing interest in the use of sub-Tenon's blocks utilizing a blunt cannula 1-5.

Even with the use of blunt canulae sub-Tenon's block, serious problems can still occur, especially in myopic patients with large axial length. In phakic IOL surgery,topical anesthesia has been used successfully for years. Topical anesthesia has several advantages over regional infiltrative techniques, the foremost of which is the abolition of any risk of inadvertent injury of the globe or orbital contents 6,7,8. It has a high rate of patient satisfaction, but still there are some patients that experience intraoperative discomfort.

In this study we compared topical anesthesia alone with topical anesthesia plus intracameral lidocaine 1% in patients undergoing posterior chamber phakic intra ocular lens;Vision implantable collamer lens ( ICL/toric ICL) surgery.Intracameral anesthesia is a common adjunct to topical anesthesia in anterior segment surgery9. It probably provides sensory blockage of the iris and ciliary body and thereby relieves discomfort experienced during IOL placement. Intracameral lidocaine alone dilates the pupil well 10 and this is believed to be because of the direct action of lidocaine on the iris, which in turn causes muscle relaxation.

DETAILED DESCRIPTION:
were enrolled in this study after obtaining approval from the institutional ethical committee and written patients consent. We estimated our sample size based on a method described by Lerman. A sample size of 45 will detect a 20% difference between each group; this will give an alpha value of 0.05 with a power of 80%. With a fall-out rate of approximately 19%, we decided to increase the number of patients in each group to 51.All patients were assessed and only those who were deemed suitable for topical and intracameral lidocaine 1% were included in the study.Very anxious patients were omitted from the study.

We are planning a study of matched sets of patients receiving the experimental and control treatments with 1 matched control(s) per experimental subject. Prior data indicate that the probability of a treatment failure among controls is 0.05 and the correlation coefficient for exposure between matched experimental and control subjects are 0.1. If the true odds ratio for failure in experimental subjects relative to control subjects is 0.1, we will need to study 51 experimental subjects with 1 matched control(s) per experimental subject to be able to reject the null hypothesis that this odds ratio equals 1 with probability (power) 0.7. The Type I error probability associated with this test of this null hypothesis is 0.3.

All the operations were done by one surgeon (SE).Patients were prepared for bilateral ICL/TICL procedure on the same day.Group I (1 eye) received topical anesthetic drops and Group 2 (the second eye) received topical anesthesia plus intracameral lidocaine 1% at the start of sugery through the 3.00 mm corneal incision. Before giving the anesthetics, a peripheral vein was cannulated and heart rate, oxygen saturation and non-invasive arterial blood pressure were monitored.Topical anesthesia was done with 2% tetracaine local anesthetic drops .

Pain was estimated by the patient using a simple pain score: no pain =0; that does not interfere with the surgical technique, discomfort=1; the surgical technique is performed with difficulty, pain=2; the surgeon is unable to continue the surgical technique. The scoring was done during different stages of surgery: lid retraction while inserting a speculum, tolerance to the microscope light, corneal incision, intraocular lens insertion, tucking of footplates, irrigation and aspiration (I/A) of viscoelastic, and peripheral iridectomy. The surgical technique was performed through a clear corneal 3.0 mm tunnel incision, followed by sodium hyaluronate injection, ICL/toricICL implantation(V4B,STAAR,California,USA) and unfolding, tucking of trailing footplates then side port incision and tucking of leading footplates, MIOSTAT 0.01% (Alcon,Texas,USA) injection, then peripheral iridectomy .

ELIGIBILITY:
Inclusion Criteria:

* any age
* calm patient
* agreed

Exclusion Criteria:

* co agulopathy anxious refusal

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
PAIN | 15 MINUTES

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Ali, Lecturer, Principal Investigator — Cairo University
Locations (1):
- Magrabi Aseer ,KSA, Khamis Mushait, West, Saudi Arabia